CLINICAL TRIAL: NCT01952210
Title: The Effectiveness of a Nutritional Consultation and Exercise Program in Esophageal Cancer Patient Receiving Neoadjuvant Chemoradiation.
Brief Title: Effectiveness of a Nutritional Consultation and Exercise Program in Esophageal Cancer Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201205017RIC
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutrition consultation and exercise program (Experimental): individual nutritional consultation and exercise
  Interventions: Behavioral: nutritional consultation and exercise program
- usual care (Active Comparator): pre-CCRT education included self-care during CCRT and body weight maintenance
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: nutritional consultation and exercise program — The protocol involved 20-30 minutes of individual-based nutrition consultation every week during the 8-week chemoradiation therapy. The exercise program consisted of upper extremity muscle training and walking exercise at 45%-65% of maximal heart rate reserve, 3 times per week, 20-30 minutes per session.
  Other Names: nutritional consultation
  Arms: nutrition consultation and exercise program
Behavioral: usual care — pre-CCRT education included self-care during CCRT and body weight maintenance
  Other Names: pre-CCRT education
  Arms: usual care

SUMMARY:
In this randomized pilot study, a nutritional consultation combining exercise program is planned for 25 locally advanced esophageal cancer patients undergoing neoadjuvant chemoradiation. The purpose of this study is to determine the effects of nutritional and exercise intervention in locally advanced esophageal cancer patients undergoing neoadjuvant chemoradiation.

DETAILED DESCRIPTION:
Patients with esophageal cancer are often malnourished at presentation due to the primary symptom of dysphagia. Treatments for esophageal cancer are commonly multimodal, incorporating polychemotherapy, radiotherapy and surgery. These treatments frequently cause or exacerbate poor nutritional status. Recent literature has proved that malnutrition is associated with longer hospital stays, reduced responses to and increased complications from therapies, increased costs, worse quality of life and lower survival rate. The aim of this study was to investigate the effectiveness of an intensive nutritional consultation and exercise program on nutritional status and outcomes in patients undergoing chemoradiation for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of locally advanced esophageal cancer, neoadjuvant chemoradiation is indicated
* Informed consent signed

Exclusion Criteria:

* stage IV, underwent palliative chemotherapy or radiotherapy patient
* clinically significant cardiac or pulmonary disease
* Unable to walk or exercise

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
General nutritional status | 10 weeks
  Measure tools included patient-generated-subjective global assessment score, hand-grip strength, body weight, body composition analysis, and 6-mim walk test were used to define the general nutritional status of esophageal cancer patient. The study measures were chosen on the basis that they had been utilized in previous cancer trials examining the effects of various interventions on weight loss, endurance and strength, and simple enough to be administered in the clinical setting.

SECONDARY OUTCOMES:
Treatment tolerance | 10 weeks
  To evaluate the treatment tolerance, the following data were assessed: number of treatment breaks or delay for toxicity, grading of acute chemoradiation-related toxicity, number of unplanned hospitalization for adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chia-Hui Chen, Principal Investigator — Department of Nursing, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan